CLINICAL TRIAL: NCT03958253
Title: I-STEP: Increasing Screening Through Engaging Primary Care Providers
Brief Title: Lung Cancer Screening Protocol
Acronym: I-STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: BJC HealthCare, Barnes-Jewish St. Peters Hospital (Unknown); Decatur Memorial Hospital (Unknown); Memorial Health System (Other); Sarah Bush Lincoln Health System (Unknown); Southern Illinois Healthcare (Unknown); Cox Health Systems (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 201811093
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Lung Cancer Screening

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge cluster randomized trial in which the intervention condition (toolbox) is sequentially assigned to participating hospitals (screening centers) in 6 clusters at different time-delays and where pre-intervention data serves as the control. By the end of the study, all clusters have been exposed to the intervention and each cluster has provided data for the control and intervention conditions. Independent samples of primary care providers are enrolled at each period within a cluster, thus, it is a repeated cross-sectional study. The order of the entry into the intervention phase is randomized based on levels of readiness
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung Cancer Screening Toolbox (Experimental): * WU Staff will train local screening staff using a train-the-trainer model three months prior to the intervention and will provide technical assistance on an ongoing basis.
  * During the 3 hour train-the-trainer session, the selected staff from the referral sites will learn about the program, receive an orientation to the toolbox elements, and discuss how to adapt the elements of the toolbox to their referral sites.
  Interventions: Other: Toolbox for Lung Cancer Screening

INTERVENTIONS:
Other: Toolbox for Lung Cancer Screening — -Toolbox of evidence-based elements that a primary care or referral site could implement to address known barriers to screening and referral, as well as required elements for screening. These elements will be designed to be adaptable to the unique needs and screening processes of the participating practices.
  * Patient education materials
  * Primary care practice educational materials
  * Pack-years/eligibility calculator
  * Local referral process guide
  * Smoking cessation materials and support
  * Shared decision-making guide
  * LDCT best practice guidelines

SUMMARY:
The successful implementation of lung cancer screening across diverse setting requires working with the community and primary care practices. Collaborating across diverse community-based sites will employ local knowledge and culture in the understanding of the health problem and identifying and implementing solutions that are appropriate for all partners (patients, primary care, referral centers). Enhanced, culturally-competent communication with patients at high risk for lung cancer can narrow inequities in screening awareness, referral, and utilization, as well as improve lung cancer outcomes across diverse patients and communities. Promoting partnerships among physicians, staff, and patients; creating routines; and tailoring materials to each clinician's situation have been show to increase the proportion of patients receiving screening.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in the trial, screening centers have to be existing members of the BJC Collaborative.
* Primary Care Providers have to have a referral relationship with the screening center; serve adult patients who may be screening-eligible, and are willing to interact with the referral site to implement referral for LDCT.

Exclusion Criteria:

There are not any exclusion criteria for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Number of initial low-dose CT (LDCT) scan screenings per month per screening center | Completion of study (estimated to be 21 months)
  -Screening will be defined as completed initial screen for lung cancer

SECONDARY OUTCOMES:
Number of primary care providers who refer at least two patients per month for LDCT | Completion of study (estimated to be 21 months)
Percent of patients referred who are screen-eligible | Completion of study (estimated to be 21 months)
  Defined as the number of screen-eligible patients divided by the total of screening procedures performed
Percent of patients referred who complete screening | Completion of study (estimated to be 21 months)
  Defined as the number of patients referred for screening divided by the total number of screening procedures performed.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee S James, Ph.D., MPH, Principal Investigator — Washington University School of Medicine; Graham A Colditz, M.D., DrPH, Principal Investigator — Washington University School of Medicine
Locations (7):
- United States (7):
  - Southern Illinois Healthcare, Carbondale, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Sarah Bush Lincoln Health System, Mattoon, Illinois
  - Memorial Health System, Springfield, Illinois
  - BJC HealthCare, Barnes-Jewish St. Peters Hospital, City of Saint Peters, Missouri
  - CoxHealth, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Practice level and screening center aggregate numbers may be made available to investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning in 3 months and ending 5 years following article publication
Access Criteria: Proposals should be directed to aimeejames@wustl.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Salazar AS, Sekhon S, Rohatgi KW, Nuako A, Liu J, Harriss C, Brennan E, LaBeau D, Abdalla I, Schulze C, Muenks J, Overlot D, Higgins JA, Jones LS, Swick C, Goings S, Badiu J, Walker J, Colditz GA, James AS. A stepped-wedge randomized trial protocol of a community intervention for increasing lung screening through engaging primary care providers (I-STEP). Contemp Clin Trials. 2020 Apr;91:105991. doi: 10.1016/j.cct.2020.105991. Epub 2020 Mar 14. PMID 32184197
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu